CLINICAL TRIAL: NCT03601416
Title: Intravenous Human Umbilical-Cord-Derived Mesenchymal Stem Cells For Moderate and Severe Bronchopulmonary Dysplasias in Children
Brief Title: Human Mesenchymal Stem Cells For Moderate and Severe Bronchopulmonary Dysplasia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xia Yunqiu, doctor, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Xia Yunqiu
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: human umbilical cord -derived mesenchymal stem cells; moderate and severe bronchopulmonary dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transplantation of Mesenchymal Stem Cell (Experimental): Mesenchymal stem cell will be given to participants with moderate and severe bronchopulmonary dysplasia.
  Interventions: Drug: Transplantation of mesenchymal stem cell
- No Transplantation of Mesenchymal Stem Cell (Active Comparator): Mesenchymal stem cell will be not given to participants with moderate and severe bronchopulmonary dysplasia.
  Interventions: Drug: No Transplantation of Mesenchymal Stem Cell

INTERVENTIONS:
Drug: Transplantation of mesenchymal stem cell — Human umbilical cord-derived mesenchymal stem cell will be given to participants through intravenous infusion.
  Dose A - 1 million cells per kg Dose B - 5 million cells per kg
  Arms: Transplantation of Mesenchymal Stem Cell
Drug: No Transplantation of Mesenchymal Stem Cell — Human umbilical cord-derived mesenchymal stem cell will be not given to participants through intravenous infusion.
  Arms: No Transplantation of Mesenchymal Stem Cell

SUMMARY:
This study is an open-label, single-center, dose escalation study to evaluate of safety and efficacy of human umbilical cord -derived mesenchymal stem cells (hUC-MSCs) in children with moderate and severe bronchopulmonary dysplasia.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) is one of the most common chronic lung diseases with poor prognosis, especially in preterm infants with moderate and severe BPD. However, there is lack of effective therapies for this disease.

hUC-MSCs are widely used in clinic due to their low immunogenicity and convenient to get.Many animal study had shown that hUC-MSCs had therapeutic effects on a variety of animal models of lung disease.Furthermore,there are a large number of clinical trials of MSCs applied to various system diseases and the safety was verified.So,the main purpose of this study is to evaluate the safety and efficacy of hUC-MSCs in participants with moderate and severe bronchopulmonary dysplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with moderate and severe bronchopulmonary dysplasia are not well treated by routine therapy
2. The legal representative or the participant had signed consent.

Exclusion Criteria:

* 1. Severe underlying diseases (e.g. systemic and hematological malignancies, heart failure, liver and kidney failure, immune deficiency, severe infectious diseases, III-IV grade pulmonary hypertension, Lung transplantation, current indications of acute surgery after lung transplantation) 2. Participants whose age is more than 1 year old.

Ages: 28 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the accumulative duration of oxygen therapy | from the time of diagnosis to the time of stopping oxygen therapy
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for moderate and severe bronchopulmonary dysplasia.

SECONDARY OUTCOMES:
Changes of blood pressure in participants | 24 hours after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for moderate and severe bronchopulmonary dysplasia. Blood pressure is measured by electronic sphygmomanometer .
Changes of heart rate in participants | 24 hours after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for moderate and severe bronchopulmonary dysplasia.

OTHER OUTCOMES:
Changes of respiratory rate in participants | 24 hours after administration
  To evaluate the safety of human umbilical cord -derived mesenchymal stem cells for moderate and severe bronchopulmonary dysplasia.
Changes of high-resolution chest CT in participants | within 2 years after administration
  To evaluate the safety and efficacy of human umbilical cord -derived mesenchymal stem cells for moderate and severe bronchopulmonary dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Fu, Study Chair — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn SY, Chang YS, Kim JH, Sung SI, Park WS. Two-Year Follow-Up Outcomes of Premature Infants Enrolled in the Phase I Trial of Mesenchymal Stem Cells Transplantation for Bronchopulmonary Dysplasia. J Pediatr. 2017 Jun;185:49-54.e2. doi: 10.1016/j.jpeds.2017.02.061. Epub 2017 Mar 21. PMID 28341525
- [Background] Laube M, Stolzing A, Thome UH, Fabian C. Therapeutic potential of mesenchymal stem cells for pulmonary complications associated with preterm birth. Int J Biochem Cell Biol. 2016 May;74:18-32. doi: 10.1016/j.biocel.2016.02.023. Epub 2016 Feb 27. PMID 26928452
- [Background] Hansmann G, Fernandez-Gonzalez A, Aslam M, Vitali SH, Martin T, Mitsialis SA, Kourembanas S. Mesenchymal stem cell-mediated reversal of bronchopulmonary dysplasia and associated pulmonary hypertension. Pulm Circ. 2012 Apr-Jun;2(2):170-81. doi: 10.4103/2045-8932.97603. PMID 22837858
- [Derived] Wu X, Xia Y, Zhou O, Song Y, Zhang X, Tian D, Li Q, Shu C, Liu E, Yuan X, He L, Liu C, Li J, Liang X, Yang K, Fu Z, Zou L, Bao L, Dai J. Allogeneic human umbilical cord-derived mesenchymal stem cells for severe bronchopulmonary dysplasia in children: study protocol for a randomized controlled trial (MSC-BPD trial). Trials. 2020 Jan 31;21(1):125. doi: 10.1186/s13063-019-3935-x. PMID 32005282